CLINICAL TRIAL: NCT07097402
Title: Examination of a Self-Compassion Course for Healthcare Providers Working With People With Multiple Sclerosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Simpson (Other)
Responsible Party: Sponsor-Investigator, Robert Simpson, Principal Investigator, University of Toronto
Organization: University of Toronto (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2072
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Burnout; Compassion
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-compassion course (Experimental): 6-week manualized online Self-Compassion for Healthcare Communities course
  Interventions: Behavioral: Self-compassion intervention (Self-Compassion for Healthcare Communities course)

INTERVENTIONS:
Behavioral: Self-compassion intervention (Self-Compassion for Healthcare Communities course) — An online 6-week mindful self-compassion course with weekly sessions.

SUMMARY:
Clinical staff working with people with multiple sclerosis often face emotional fatigue and high levels of burnout. The Self-Compassion for Healthcare Communities course is an evidence-based intervention that teaches participants how to meet distress with kindness and care. This study will recruit up to 40 staff from the Barlo MS Clinic at St. Michael's Hospital to take part in a 6-week, 6-session Self-Compassion for Healthcare Communities course. Participants will be asked to complete surveys before and after the course to understand the effects of the course on a range of outcomes. Participants will be invited to take part in one qualitative interview on their perspectives on the course.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older
2. Able to understand spoken and written English
3. Current professional affiliation with the Barlo MS clinic

Exclusion Criteria:

1) Severe active mental health impairment (psychosis, suicidality)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment | 6 months
  The investigators will measure the number of participants eligible for and recruited to the study.
Retention | 6 months
  The investigators will measure the percentage of participants who complete outcome data.
Adherence | 6 months
  The investigators will measure the number of participants who completed the Self-Compassion for Healthcare Communities course.
Follow-up rates | 6 months
  The investigators will measure the percentage of participants who complete outcome measures pre-intervention, post-intervention, and at 3 months post-intervention.

SECONDARY OUTCOMES:
Professional Quality of Life Scale (ProQOL) Version 5 | Baseline, post-intervention (6 weeks after baseline), and 3 months post-intervention
  Measures the positive and negative effects of one's compassion for those that they help. Includes with subscales for compassion satisfaction and compassion fatigue (including burnout). Answers are assessed using a 5-point Likert scale, with higher scores on the compassion satisfaction sub-scale indicating higher compassion satisfaction, and higher scores on compassion fatigue sub-scale indicating higher burnout.
Self-Compassion Scale - Short Form | Baseline, post-intervention (6 weeks after baseline), and 3 months post-intervention
  Measures how one typically acts towards themselves in difficult times. The total score ranges from a 1-5, with higher scores representing high self-compassion.
Relational Compassion Scale | Baseline, post-intervention (6 weeks after baseline), and 3 months post-intervention
  Measure's ones tendencies for receiving and providing relational compassion. Answers are assessed using a 4-point Likert scale. Higher scores represent higher compassion for self and others.
Perceived Stress Scale-10 | Baseline, post-intervention (6 weeks after baseline), and 3 months post-intervention
  Measures one's thoughts and feelings pertaining to stress. The total score can range from 0-40, with higher scores indicating higher perceived stress.
Difficulties in Emotion Regulation Scale - Short Form | Baseline, post-intervention (6 weeks after baseline), and 3 months post-intervention
  Measures emotion regulation. Answers are assessed using a 5-point Likert scale. Higher values indicate greater difficulties in emotion regulation.
Dispositional Joy Scale | Baseline, post-intervention (6 weeks after baseline), and 3 months post-intervention
  Measures trait/dispositional joy. Answers are assessed using a 7-point Likert scale, with higher scores representing higher joy.

CONTACTS AND LOCATIONS:
Locations (1):
- Unity Health Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No